CLINICAL TRIAL: NCT02762045
Title: Phase I Clinical Trial of Recombinant Adenovirus Type 5 Therapeutic AIDS Vaccine Expressing Gag
Brief Title: Clinical Trial of Recombinant Adenovirus Type 5 AIDS Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Beijing Ditan Hospital (Other); National Institutes for Food and Drug Control, China (Other)
Responsible Party: Principal Investigator, Yi Zeng, Yi Zeng, Departement Director, Centers for Disease Control and Prevention, China, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDCPChina
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Therapeutic Vaccine HIV Adenovirus type 5 vector
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose Ad5-gag or Placebo (Experimental): 1ml low dose Ad5-gag(2x10^9VP) or Preservation solution at weeks 0 and weeks 4.
  Interventions: Biological: Ad5-gag; Biological: Placebo
- Medium dose Ad5-gag or Placebo (Experimental): 1ml medium dose Ad5-gag(2x10^10VP) or Preservation solution at weeks 0 and weeks 4.
  Interventions: Biological: Ad5-gag; Biological: Placebo
- High dose Ad5-gag or Placebo (Experimental): 1ml high dose Ad5-gag(2x10^11VP) or Preservation solution at weeks 0 and weeks 4.
  Interventions: Biological: Ad5-gag; Biological: Placebo

INTERVENTIONS:
Biological: Ad5-gag — Ad5-gag is used as vaccine in all arms.
Biological: Placebo — Preservation Solution is used as control in all arms.
  Other Names: Preservation Solution

SUMMARY:
This is a randomized, double-blind placebo-controlled dose-escalation clinical trial to evaluate the safety and the immunogenicity of Adenoviral vector 5 HIV-1 vaccines in subjects receiving stable highly active antiretroviral therapy(HAART) .

DETAILED DESCRIPTION:
Patients continue antiretroviral medications throughout the course of this study. Three groups of patients receive dose-escalation (2×10^9VP, 2×10^10VP or 2×10^11VP) injections of Adenovirus vector vaccine (Ad5-gag). Two weeks post immunization of lower dose, if the vaccine is safe and well tolerant, the next dose of immunization will begin. patients are monitored for safety 72 hours after each immunization. In addition, each patient records adverse events in a diary. Patients have regular physical exams, pregnancy tests, and blood drawn for virologic and immunologic assessments. The induction of HIV-specific responses will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Are willing to participate this study and available for follow-up for the duration of the study.
* Men and women aged 18-50 years.
* Are HIV-positive.
* Have been taking stable anti-HIV drugs for at least 6 months.
* CD4 count ≥ 350 cells/mm3
* Plasma viral load < 50 copies/ml.
* Willing to use acceptable forms of contraception at least 21 days prior to first vaccination until 56 days after the last vaccination.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* History of previous vaccination with an HIV-1 vaccine.
* Use of immunoinhibitory agents, such as corticosteroids or cytotoxic drugs by oral administration, injection route or inhalation route within 6 months of study entry (But corticosteroids used for allergic rhinitis and skin topical application of corticosteroids were not included); Use of immunomodulatory agents including but not limited to interleukin-2(IL-2） and granulocyte-macrophage colony-stimulating factor (GM-CSF) within 30 days of study entry.
* Use of blood products within 3 months of study entry.
* Use of other experimental drugs within 3 months of study entry.
* Any immunization within 3 months of study entry.
* Comply with any of the following items： Active pulmonary tuberculosis； History of serious adverse reaction to other vaccines； Serious asthma； Have untreated thyroid disease; Syphilis
* Laboratory values（Comply with any of the following items）:

Hemoglobin < 100 g/L (male subjects)，<90 g/L (female subjects)； Absolute neutrophil count ≤ 1000 cells/mm3； Serum creatinine ≥15 mg/L，endogenous creatinine clearance rate <50 ml/min； alanine aminotransferase（ALT）, aspartate aminotransferase(AST) ≥3× upper limit of normal range； Total bilirubin ≥2× upper limit of normal range

* Clinically significant electrocardiogram changes.
* Hypertension ( If it is well controlled by medication and is less than 150/100mmHg , should not be excluded) and other cardiac disease；
* Any medical, psychiatric, social condition, occupational reason judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of local and systemic adverse events | 12 months
  To evaluate the safety and tolerance of a replication defective adenovirus expressing HIV-1 gag in HIV-1 infected subjects on highly active antiretroviral therapy.

SECONDARY OUTCOMES:
Immunogenicity of vaccine | 24 month
  To evaluate immune responses pre- and post-immunization and between the vaccine and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zeng, M.D., Study Director — National Institute for Viral Disease Control and Prevention, China CDC; Xia Feng, M.D. Ph.D, Principal Investigator — National Institute for Viral Disease Control and Prevention, China CDC; Ke Xu, Ph.D, Principal Investigator — National Institute for Viral Disease Control and Prevention, China CDC
Locations (1):
- Beijing Ditan Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided